CLINICAL TRIAL: NCT01775644
Title: Avastin ® First Line and Where Applicable Beyond First Progression With Metastatic Colorectal Carcinoma
Brief Title: An Observational Study of Avastin in Participants With Metastatic Colorectal Cancer (KORALLE)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28120
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Metastatic Colorectal Cancer Participants: Administration of treatment will be as used in normal daily routine under local labelling in 4 subgroups- participants with liver and/or lung metastases, potentially resectable after a response to a systemic therapy and clinically operable; participants with tumor related symptoms, risks for complications or fast progression for whom quick proliferation control is needed; "asymptomatic" participants (indolent tumor) without the option of a metastases resection (no pressure for remission) for whom the aim of the therapy is proliferation control and participants without classification.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Administration of treatment will be as used in normal daily routine under local labeling.
  Other Names: Avastin

SUMMARY:
This observational multicenter study will evaluate the differences in progression-free survival defined in specific subgroups of participants with metastatic colorectal cancer receiving bevacizumab (Avastin). Further, safety and efficacy in daily routine will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Participants with metastatic colorectal cancer where physician has decided to give a first-line, fluoro-pyrimidine-based combination therapy with bevacizumab according to Summary of Product Characteristics (SmPC)

Exclusion Criteria:

* Contraindications for bevacizumab according to SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with metastatic colorectal cancer
Sampling Method: Probability Sample
Enrollment: 3003 (Actual)
Dates: Start 2012-12-14 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
Median Progression-Free Survival Time in Defined Participant Subgroups as Assessed by Response Evaluation Criteria In Solid Tumors (RECIST) | Baseline up to 5 years

SECONDARY OUTCOMES:
Percentage of Participants by Prognostic Factors | Baseline up to 5 years
Percentage of Participants by Carcinoembryonic Antigen Tumor Marker | Baseline
Percentage of Participants by Cancer Antigen 19-9 Tumor Marker | Baseline
Percentage of Participants by Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline
Percentage of Participants by Comorbidity Index as per Carlson Method | Baseline
Percentage of Participants by RAS Mutation Status | Baseline
Percentage of Participants by Cancer Metastasation Status | Baseline
Percentage of Participants According to Previous Treatment Regimen of Bevacizumab | Baseline
Progression-Free Survival as Assessed by RECIST (Overall) | Baseline up to 5 years
Overall Survival in Daily Routine Practice | Baseline up to 5 years
Overall Survival in Defined Participant Subgroups in Daily Routine Practice | Baseline up to 5 years
Percentage of Participants Showing Overall Response in Daily Routine Practice as Assessed by RECIST | Baseline up to 5 years
Number of Treatment Application Schemes of Bevacizumab Daily Routine Practice | Baseline up to 5 years
Number of Participants With Adverse Event | Baseline up to 5 years
Number of Participants With Reason for Bevacizumab Treatment Modifications and Discontinuation in Defined Participant Subgroups | Baseline up to 5 years
Total Cumulative Therapy Dose of Bevacizumab | Baseline up to 5 years
Percentage of Participants With Treatment Success | Baseline up to 5 years
Percentage of Participants With Resection | Baseline up to 5 years
Number of Physicians Satisfied With Treatment | Baseline up to 5 years
Percentage of Participants Without Resection by Reason | Baseline up to 5 years
Percentage of Participants With Follow-Up therapy | Baseline up to 5 years
Percentage of Participants in Defined Participant Subgroups Showing Overall Response in Daily Routine Practice as Assessed by RECIST | Baseline up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche